CLINICAL TRIAL: NCT01543646
Title: Rapid Imaging Assessment of the Liver Using Multiparametric Magnetic Resonance
Brief Title: Multiparametric MR for Rapid Imaging Assessment of the Liver
Acronym: RIAL
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Oxford (Other)
Collaborators: British Heart Foundation (Other); Oxford University Hospitals NHS Trust (Other)
Responsible Party: Sponsor
Other Study IDs: RIAL MR
Record Dates: First submitted 2012-02-13; First posted 2012-03-05 (Estimated); Last update posted 2012-03-05 (Estimated); Status verified 2012-03

CONDITIONS: Liver Cirrhosis; Fatty Liver
Keywords: Hepatology; Liver Cirrhosis; Fatty Liver
MeSH Terms: conditions — Liver Cirrhosis; Fatty Liver

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Fresh frozen plasma, frozen serum, and whole blood for DNA analysis
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Liver Biopsy patients: All patients due to have a liver biopsy for the assessment of parenchymal liver disease.

SUMMARY:
The RIAL study aims to investigate whether non-invasive measurement of liver fat, iron content and fibrosis are as accurate as liver biopsy specimens in determining if patients have non-alcoholic fatty liver disease (NAFLD) or steatohepatitis (NASH), or other suspected liver disease.

Currently, the gold-standard for the diagnosis and staging of liver disease is a liver biopsy.

In this study, consecutive patients will be offered a multiparametric MR scan to assess their liver while they await a liver biopsy.

Study time-frame: The scan will be performed in the 6-week period before their biopsy, and results will be compared to biopsy findings. results will be presented at the end of the study when MR data outcomes are compared to gold-standard biopsy dat. Participants will only have to attend one study visit to participate - there will be no patient follow-up.

DETAILED DESCRIPTION:
Obesity per se as a cause of liver dysfunction and failure has been well studied. However, although it is a very common disease, at present the only reliable way to diagnose it is with percutaneous liver biopsy. This is painful and not without risk, as the liver is a highly vascular organ. Even with ultrasound guidance, it is still a diagnostic test that is underused as it carries a 1:1000 risk of serious adverse events (eg bleeding, infection, bowel perforation) because it is invasive. Moreover, the patients requiring the test often have impaired clotting of their blood due to liver dysfunction, and so are at higher risk of bleeding, and need to be observed in hospital for a few hours after the procedure. This adds to the cost of the procedure. As a result of these factors, liver biopsy is not used in all patients for whom NAFLD, NASH or other liver disease are suspected, unless the patients have clinically moderate to severe disease.

With the increasing prevalence of obesity in the community, NASH and NAFLD are becoming increasingly common, and there is a need for a reliable, feasible and cost-effective non-invasive diagnostic tool for these conditions. Moreover, they often coexist with other liver diseases (eg tumours, or autoimmune liver disease). There are approximately 1.5million UK adults with mild to moderate liver disease which, at present, cannot be ascertained non-invasively.

Developments in magnetic resonance medicine may allow us to accurately diagnose liver fibrosis, using the amount of extracellular fluid (ECF) as a biomarker for fibrosis. T1 mapping of the liver can reliably show differences in ECF content and thereby allow quantification of the degree of liver fibrosis. In conjunction with MR spectroscopy and T2* mapping for concurrent interpretation of lipid and iron content, this will allow rapid non-invasive diagnosis of the type and/or severity of many common liver diseases (NAFLD/NASH, hepatitis, iron overload).

ELIGIBILITY:
Inclusion Criteria:

* Male or Female over 18 years of age due for diagnostic liver biopsy
* Participant is willing and able to give informed consent for participation in the study.

Exclusion Criteria:

* Any contraindication to magnetic resonance imaging (inc pregnancy, extensive tattoos, pacemaker, shrapnel injury, severe claustrophobia).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study aims to recruit 60 patients due to undergo liver biopsy to establish a diagnosis of liver disease. These patients will be recruited from the Oxford Radcliffe Hospitals clinics by Dr Jane Collier, consultant hepatologist, and her colleagues. Each patient will be scheduled for an ultrasound-guided liver biopsy as part of their usual care. We will ask these patients if they wish to take part in our research study, and offer to arrange the research scans before the biopsy and a time of their choice.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2011-03; Primary Completion 2012-09 (Estimated); Study Completion 2012-09 (Estimated)

PRIMARY OUTCOMES:
Liver fat content | Day 1
  Liver fat content in this study is measured with MR spectroscopy during cardiac-gated breatholds
Liver fibrosis | Day 1
  Liver fibrosis is measured by the T1 relaxation time in milliseconds (continuous variable) using MR. Higher degrees of fibrosis are predicted to have a higher T1 value. These results will be compared to gold-standard histology.

CONTACTS AND LOCATIONS:
Overall Officials: Eleanor Barnes, BSc MBBS PhD, Study Director — University of Oxford; Stefan Neubauer, MD, Study Director — University of Oxford
Locations (1):
- John Radcliffe Hospital, Oxford University Hospitals NHS Trust, Oxford, England, United Kingdom

REFERENCES:
- [Derived] Dennis A, Kelly MD, Fernandes C, Mouchti S, Fallowfield JA, Hirschfield G, Pavlides M, Harrison S, Chakravarthy MV, Banerjee R, Sanyal A. Correlations Between MRI Biomarkers PDFF and cT1 With Histopathological Features of Non-Alcoholic Steatohepatitis. Front Endocrinol (Lausanne). 2021 Jan 27;11:575843. doi: 10.3389/fendo.2020.575843. eCollection 2020. PMID 33584535